CLINICAL TRIAL: NCT05577546
Title: The Effect of Conservative Treatment on Gait Biomechanics in Adolescent Idiopathic Scoliosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: University of Ljubljana (Other); Moor Orthotics and Prosthetics (Unknown)
Responsible Party: Principal Investigator, Ahsen Büyükaslan, Ahsen Buyukaslan, PT, PhD(c), Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUET2020-798
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Idiopathic Scoliosis; Gait Disorder, Sensorimotor
Keywords: adolescent idiopathic scoliosis; gait analysis; gait biomechanics; kinetic; kinematic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brace group (Experimental): Fifteen patients with AIS will be included in this group. The scoliosis brace, whose characteristics are described below under the "Brace" heading, will be worn by the patient for 12 weeks. Although the daily brace wearing time varies between 20-23 hours, depending on the patient, it will be determined according to the physician's recommendation. Compliance regarding the brace will be monitored from the parent-controlled charts where the daily wearing time is recorded by the patient
  Interventions: Other: Moor S brace treatment
- Brace and Schroth exercise group (Experimental): Fifteen patients with AIS will be included in this group, they will be treated by brace and exercise during 12 weeks. The same brace treatment protocol as the brace group will be applied for this group. Additionally, Schroth Three-Dimensional Scoliosis Exercise Treatment will be applied to this group by the researcher physiotherapist at the brace center. Exercise therapy will be carried out at the brace center once a week with the researcher physiotherapist, and 45 min a day, 4 days a week in the form of home exercises. The number of exercise sets and repetitions will be determined by the researcher physiotherapist according to the patient, considering deformity severity and flexibility, generalized joint hypermobility, bone maturation, menarche status and the risk of progression. Compliance with the home exercise program (frequency and duration) will be recorded by the patients in a home exercise diary for 12 weeks.
  Interventions: Other: Moor S brace treatment; Other: Schroth Three-Dimensional Scoliosis Exercise Treatment
- Healthy control group (No Intervention): Fifteen healthy volunteers between the ages of 10-18 will be included in this group. No intervention will be applied to this group and they will only be assessed, and their findings obtained from the gait analysis will compare with the patient groups.

INTERVENTIONS:
Other: Moor S brace treatment — The rigid MOOR-S Brace controls the thoracic, lumbar and pelvis blocks very tightly, is modelled and produced according to deformity type and patients body size considering the standardization of the MOOR-S Model. It is a CAD-CAM design-based rigid torocolumbosacral orthosis, using polypropylene material, which is opened from the front, and tightness can be adjusted by the patients with the help of straps. Additional corrective forces can be applied with pads that can be added to the brace. The amount of corrective forces in the MOOR-S brace is decided by the experienced orthotist, taking into account risk of progression, the flexibility of the spine deformity, Cobb angle, bone maturation and age. An external stimulus is provided that directs the protracted shoulder to slightly to the posterior by the shoulder part, located on the anterosuperior side of the brace.
  Arms: Brace and Schroth exercise group; Brace group
Other: Schroth Three-Dimensional Scoliosis Exercise Treatment — Schroth Three-Dimensional Scoliosis Exercise Treatment has the main features of physiotherapeutic scoliosis-specific exercises: 1) Three-dimensional self-correction, 2) Training activities of daily living (ADL), and 3) Stabilization of the corrected posture. The basic principles of the Schroth method are autoelongation, deflection, derotation, rotational angular breathing and stabilization. Exercise therapy will be carried out at the brace center once a week with the researcher, and 45 min a day, 4 days a week in the form of home exercises. The number of exercise sets and repetitions will be determined by the physiotherapist according to the patient, considering deformity severity and flexibility, generalized joint hypermobility, bone maturation, menarche status and the risk of progression. Compliance with the home exercise program (frequency and duration) will be recorded by the patients in a home exercise diary for 12 weeks.
  Other Names: Schroth Therapy
  Arms: Brace and Schroth exercise group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional complex progressive structural deformity of the growing spine. Asymmetric changes in both the anatomical structure and strength of the muscles due to deformity affect weight distribution and joint moments in the trunk and lower extremities. As the spine transfers loads through the pelvis, asymmetry in the spinal alignment creates structural or functional changes involving other parts of the kinetic chain. The deviations caused by the deformity in all three planes and the responses to it affect the kinetics and kinematics of the trunk and extremities. A number of kinetic and kinematic changes such as decreased hip muscle strength, asymmetric lateral stepping, decreased hip and pelvic joint range of motion, especially in the frontal and transverse planes, and ground reaction force asymmetry has been demonstrated in patients with AIS. Understanding the postural changes and correction strategies that affect the displacement of the center of mass, ground reaction force and center of pressure during standing and walking in adolescents with idiopathic scoliosis is fundamental to understanding the nature of the disease, disease management and guiding rehabilitation both conservative treatment and after surgery. Based on this, it was aimed to objectively measure the biomechanical effects of the forces applied to the body in the brace to control deformity and prevent progression during the growth period, to determine postural control strategies, kinetic and kinematic changes in these patients with treatment by applying MOOR-S model brace and Schroth Three-Dimensional Scoliosis Exercise Treatment as a conservative treatment method on patients with AIS. In addition, it was also aimed to determine lower extremity inequality by measuring dynamic leg length with gait analysis in individuals with functional leg length discrepancy due to scoliosis.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional complex progressive structural deformity of the growing spine. Asymmetric changes in both the anatomical structure and strength of the muscles due to deformity affect weight distribution and joint moments in the trunk and lower extremities. As the spine transfers loads through the pelvis, asymmetry in the spinal alignment creates structural or functional changes involving other parts of the kinetic chain. The deviations caused by the deformity in all three planes and the responses to it affects the kinetics and kinematics of the trunk and extremities. Various postural compensatory strategies emerge to maintain a stable position and energy conservation in deviation of the center of mass. Thorax-pelvis coordination plays an important role in maintaining the stability of the whole body in normal walking, the thorax and pelvis counter-rotate towards each other, minimizing the angular momentum of the trunk. In individuals with idiopathic scoliosis, higher in-phase and lower anti-phase coordination in the transverse planes in walking; less coordination consistency were observed in the transverse and frontal planes compared to healthy controls. Most of the studies on gait in AIS have concluded that there is no significant difference in walking speed, cadence and stride width in scoliosis patients and healthy controls. However, decreased hip and pelvic motion, increased energy consumption for gait, step pattern asymmetry, and ground reaction force asymmetry were observed in patients with AIS. A number of kinetic and kinematic changes such as decreased hip muscle strength, asymmetric lateral stepping, decreased hip and pelvic joint range of motion, especially in the frontal and transverse planes, and ground reaction force asymmetry has been demonstrated in patients with AIS. None of the studies included follow-up, most of them did not use EMG, the relationship with curvature types was not clearly revealed, and no treatment effect and follow-up results were evaluated. With this study, the deficiency in the literature will be tried to be overcome, especially in terms of the effect of conservative treatment on gait. Understanding the postural changes and correction strategies that affect the displacement of the center of mass, ground reaction force and center of pressure during standing and walking in adolescents with idiopathic scoliosis is fundamental to understanding the nature of the disease, disease management and guiding rehabilitation both conservative treatment and after surgery. Based on this, it was aimed to objectively measure the biomechanical effects of the forces applied to the body in the brace to control deformity and prevent progression during the growth period, to determine postural control strategies, kinetic and kinematic changes in these patients with treatment by applying MOOR-S model brace and Schroth Three-Dimensional Scoliosis Exercise Treatment as a conservative treatment method on patients with AIS. In addition, it was also aimed to determine lower extremity inequality by measuring dynamic leg length with gait analysis in individuals with functional leg length discrepancy due to scoliosis. Individuals who are diagnosed with AIS and decided to treat a brace, Cobb angle between 20-45 degree and age between 10-18, will be included in the study. Participants will be divided into three groups. The first group will receive MOOR-S brace treatment, the second group will receive the MOOR-S brace and Schroth Three-Dimensional Scoliosis Exercise Treatment, and the third group will not receive any intervention, this group will consist of healthy volunteers from the same age group. Full-time brace treatment will be given to the treatment groups for three months and the second group will be given a home exercise program four days a week and they will perform once a week under physiotherapist supervision. The body center of mass, ground reaction force, range of motion, joint moments and strengths, spinal flexibility, muscle activity in gait, dynamic deviation of the rotational trunk-pelvis segment position, position and orientation of the body segments in three planes, will determine statically and dynamically when they walking, it will be analyzed before and after three months treatment, patients with AIS will be compared with their healthy peers, and the effects of treatment on gait will be determined in the study sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients, diagnosed with AIS and referred to brace center for conservative treatment by the physician
* Cobb angle between of 20-45°
* ages 10 to 18 years
* no treatment before
* Individuals with family consent will be included

Exclusion Criteria:

* Spine surgery
* A history of major lower extremity trauma and associated surgery
* Leg length inequality more than 1 cm
* Other musculoskeletal pathologies that may affect gait
* Presence of transitional vertebrae
* Scoliosis due to other etiology
* Presence of infection, tumor, rheumatic and neurological disease which affected spine

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Body center of mass | Change from baseline body center of mass at 3 months
  Body center of mass and its displacement with the brace will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System (Gothenburg, Sweden), assessments will be made with the bare feet while standing and walking. Walking speed is chosen by each individual. Six walking trials will be recorded for each individual on a 15-meter walking path. The system integrated with wireless EMG (Wireless EMG system Delsys) and force platforms (AMTI) has 12 high-resolution cameras and allows the sensing of movement in three planes by Gait Module for Qualisys Track Manager software with the help of marker placed on specific anatomical reference points in the body. Instituti Orthopedici Rizzoli (IOR) Full Body marker protocol was chosen to specify anatomical landmarks.
Center of pressure | Change from baseline center of pressure at 3 months
  The Center of pressure and its displacement with the brace will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System (Gothenburg, Sweden), assessments will be made with the bare feet while standing and walking. Walking speed is chosen by each individual. Six walking trials will be recorded for each individual on a 15-meter walking path. The system integrated with wireless EMG (Wireless EMG system Delsys) and force platforms (AMTI) has 12 high-resolution cameras and allows the sensing of movement in three planes by Gait Module for Qualisys Track Manager software with the help of marker placed on specific anatomical reference points in the body. Instituti Orthopedici Rizzoli (IOR) Full Body marker protocol was chosen to specify anatomical landmarks. Markers will be placed bilaterally at points on the extremity and both sides of the body.
Thorax-pelvis coordination pattern | Change from baseline thorax-pelvis coordination pattern at 3 months
  The dynamic deviation of the rotational thorax-pelvis segment position relative to the progression line will be measured. Thorax-pelvis coordination will reveal the relative rotational range of motion between the head, pelvis and upper body in the coordinate system with the information obtained from the relevant anatomical reference points as in the literature. Thorax-pelvis coordination pattern will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System, assessments will be made with bare feet while standing and walking. The system integrated with wireless EMG and force platforms (AMTI) has 12 high-resolution cameras and allows the sensing of movement in three planes by Gait Module for Qualisys Track Manager software with the help of markers placed on specific anatomical reference points in the body.
Dynamic leg length | Change from baseline dynamic leg length at 3 months
  Dynamic leg length is the effective length of the lower limb, measured by the distance from the hip joint center to the heel, ankle joint center and forefoot, in order to determine possible functional LLD. Measuring dynamic leg length during the gait cycle takes into account the bony segmental length (foot segment, shank segment, thigh segment) and kinematic angles of the lower extremity in the sagittal, frontal and horizontal plane. Dynamic leg length will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System (Gothenburg, Sweden), assessments will be made with bare feet while standing and walking. The system integrated with wireless EMG and force platforms (AMTI) has 12 high-resolution cameras and allows the sensing of movement in three planes by Gait Module for Qualisys Track Manager software with the help of marker placed on specific anatomical reference points in the body.
Trunk, pelvis and lower extremity kinetics | Change from baseline trunk, pelvis and lower extremity kinetics at 3 months
  Using anthropometric measurements, kinematic data and ground reaction force data, joints moments and forces will be calculated with the "inverse dynamics" method. Body kinetics (kinetic analysis) includes:
  1. Ground reaction force: It will be measured in three planes as mediolateral, vertical and anteroposterior with the force platform of the system.
  2. Net moment (Nm/kg): The signals received from the muscles will be recorded by superficial EMG. As a result of the internal moment and external moment, the net moment and the flexor and extensor moment related to the dominant muscle group will be revealed.
  3. Power: The data obtained from the negative and positive mechanical power graphs will be examined concentric or eccentric contraction and power generation or absorption of the muscles.
  Body kinetics (kinetic analysis) will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System
Trunk, pelvis and lower extremity kinematics | Change from baseline trunk, pelvis and lower extremity kinematics at 3 months
  Body kinematics (kinematic analysis): The position and orientation of the relevant body segments will be measured according to the global coordinate system using the information from the markers and anthropometric data. Through kinematic analysis, joint angles of the head, trunk and extremities in three planes in different phases of gait will be measured. Body kinematics will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System (Gothenburg, Sweden), assessments will be made with bare feet while standing and walking. The system integrated with wireless EMG (Wireless EMG system Delsys) and force platforms (AMTI) has 12 high-resolution cameras and allows the sensing of movement in three planes by Gait Module for Qualisys Track Manager software with the help of marker placed on specific anatomical reference points in the body.
Time-distance parameters of gait | Change from baseline time-distance parameters of gait at 3 months
  Time-distance parameters will be measured with the data obtained from the kinematic data and force platforms.
  1. Walking speed
  2. Cadence
  3. Single and double stride length
  4. Stance and swing time
  5. Single and double support time
  6. Walk-Ratio Time-distance parameters will assess with computerized 3D gait analysis: With the optoelectronic motion capture system by Qualisys Motion Capture System (Gothenburg, Sweden), assessments will be made with bare feet while standing and walking. Walking speed is chosen by each individual. Six walking trials will be recorded for each individual on a 15-meter walking path. The system integrated with wireless EMG (Wireless EMG system Delsys) and force platforms (AMTI) has 12 high-resolution cameras and allows the sensing of movement in three planes by Gait Module for Qualisys Track Manager software with the help of marker placed on specific anatomical reference points in the body.

SECONDARY OUTCOMES:
The angle of trunk rotation | Change from baseline the angle of trunk rotation at 3 months
  The angle of trunk rotation will be measured by the scoliometer between T1-S1, and the highest value obtained in each part of the spine will be recorded. The angle of trunk rotation indicates the deviation in the transverse plane caused by vertebral rotation in that segment. The scoliometer developed by "Orthopedics Systems Incorporation®" will be used for the measurements.
Cobb angle | Baseline
  Cobb angle is the sum of upper and lower end vertebra tilt angles in standing anterioposterior radiography. The included angle of the upper vertebra endplate line with the horizontal line is measured on the imaging data and the included angle of the lower vertebra endplate line with the horizontal line is measured on the imaging data.
Risser stage | Baseline
  The Risser sign is an indirect measure of skeletal maturity, whereby the degree of ossification of the iliac apophysis by x-ray evaluation is used to judge overall skeletal development. Risser stage will be defined using patients spine radiography and physician report. Risser sign consist 5 stages. Risser 0 indicates an immature skeleton while Risser 5 indicates a mature skeleton.
Deformity classification | Baseline
  Curvature classification will be defined using patients' spine radiography and physician report. Deformity classification will be given as in the gait analysis studies in the literature, indicating a direction and localization in the form of curvature as single thoracic, single lumbar/thoracolumbar and double major
Generalised joint hypermobility | Baseline
  The presence of generalised joint hypermobility will be evaluated with the nine-point Beighton test using the cut-off ≥5 points. Evaluation consists of five parameters; the first 4 items are evaluated symmetrically in all extremities and 1 point is given for each movement that can be performed. The 5th item is evaluated as 1 point: hyperextension of the MCP joint of the fifth finger >90∘; abduction of the thumb to the forearm; elbow hyperextension >10∘; knee hyperextension >10∘; and touching the floor with the palms of the hands during trunk forward bend performed in a standing position
Health Related Quality of life | Change from baseline health related quality of life at 3 months
  Quality of life in patients with AIS will be assessed using the SRS-22 Questionnaire. SRS-22 was developed by the Scoliosis Research Society to evaluate health-related quality of life (HRQL) in patients with adolescent idiopathic scoliosis (AIS). The SRS-22 questionnaire consists of 22 items Likert type scale that allows scoring between 1-5 for each question. SRS-22 has five domains including function, pain, mental health, self-image and satisfaction. Subgroups can be evaluated separately, or the total score is obtained by summing up the scores from all questions. The total score of each section ranges from 5 to 25, only the section evaluating satisfaction from the treatment is in the range of 2-10. Scoring is obtained by dividing the total score of each section by the number of questions in that section. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Devrim Tarakcı, Assoc.Prof., Study Director — Medipol University; Janez Vodicar, Assoc.Prof., Study Director — University of Ljubljana; Ahsen Buyukaslan, PhD (c), Principal Investigator — Medipol University
Locations (1):
- University of Ljubljana, Ljubljana, Slovenia